**Document type:** Statistical Analysis Plan

Study title: Development and Pilot Test of an mHealth Interactive Education and Social Support

Intervention for Improving Postnatal Health – Phase 1

NCT number: NCT04636398

Document date: June 1, 2020

## STATISTICAL ANALYSIS PLAN - PHASE 1

The proposed research includes two separate research phases to achieve our research aims: 1) To develop optimal intervention functions and mHealth technology delivery platforms for education and peer support among postnatal women in rural India; and to pilot test the optimized intervention and assess 2) feasibility and acceptability, and 3) preliminary effectiveness on maternal and infant health outcomes. Due to the exploratory nature of these aims, the sample sizes for our two study phases have been designed for feasibility, not for adequate power for statistical testing.

**Phase 1.** Phase 1 is a developmental research phase wherein we assess women's preferences for intervention functions, processes and platforms in order to design the most appropriate intervention for full piloting.

Data collection during this phase includes capture of back-end data for participation and content, and survey (all participants) and in-depth interview (subset of participants) to understand preferences.

## Data includes:

- Backend data: intervention participation, intervention engagement, content of group discussions, content of text messaging.
- Survey: Preferences regarding group components, functions and modalities.
- In-depth interview: Preferences regarding group components, functions and modalities.

Quantitative data will be analyzed for means and proportions using STATA version 15. Text data from discussion/messaging and in-depth interviews will be analyzed for content and themes using Atlas.ti software.